CLINICAL TRIAL: NCT06667661
Title: A Home-Based Intervention to Improve Adherence to the 24-Hour Movement Guidelines in Young Children
Brief Title: A Mobile App to Improve 24-Hour Movement Guideline Adherence in Preschoolers
Acronym: Shining Star
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chelsea L. Kracht, PhD, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00160250; R00HD107158 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy; 24-Hour Movement Guidelines; Feasibility Studies; Sleep; Physical Activity; Screen Time; Sedentary Behaviors; Motor Skills; Cognition; Parent-Child Relations; Mobile Application; Health Education; Child Development
Keywords: Physical Activity; Sedentary Behavior; Sleep; Child Development; Motor Skills; Behavioral problems; Healthy; 24-Hour Movement Guidelines; Screen Time; Sedentary Behaviors; Cognition; Parent-Child Relations; Mobile Application; Health Education
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Health Education; Problem Behavior

STUDY DESIGN:
Intervention Model Description: A randomized control trial with a waitlist control design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-Week Intervention (Experimental): Participants in the intervention group will receive access to the "Shining Star" mobile health application for 12 weeks. The app provides weekly lessons and behavior-related goals focused on improving adherence to the 24-Hour Movement Guidelines (physical activity, screen time, and sleep). Parents will receive concise messages (less than 500 characters) through the app, along with links to additional resources, gamification elements, and behavior trackers. Participants and participants will also complete physical activity and sleep assessments using accelerometers and questionnaires at baseline, Week 6, and Week 12.
  Interventions: Behavioral: Shining Star mHealth App
- Wait-list Control (No Intervention): Participants in the wait-list control group will receive no intervention during the initial 12 weeks. They will complete the same assessments (physical activity, screen time, sleep, motor skills, and cognition) at baseline, Week 6, and Week 12. After the 12-week period, they will be granted access to the Shining Star mobile app and receive all lessons and resources provided to the intervention group.

INTERVENTIONS:
Behavioral: Shining Star mHealth App — The Shining Star mHealth App Intervention is a 12-week mobile health program designed to improve adherence to the 24-Hour Movement Guidelines (physical activity, screen time, and sleep) among preschool-aged children (3-4 years old). The intervention delivers weekly behavior-related goals and educational lessons to parents through a mobile app, including concise messages (<500 characters) and links to additional resources. The app also includes gamification features, behavior trackers, and a "Kids Corner" for child-friendly content. Parents receive reminders and can engage with other participants through an optional chat forum.
  Arms: 12-Week Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether a home-based mHealth intervention can improve adherence to the 24-Hour Movement Guidelines in preschool-aged children (3-4 years old) who currently meet 0 or 1 of the guidelines for physical activity, sedentary behavior, and sleep. The main questions it aims to answer are:

* Can the intervention increase the proportion of children meeting all three 24-Hour Movement Guidelines (physical activity, screen-time, and sleep)?
* Is the intervention feasible for parents to implement, as measured by a parent feedback survey?

Researchers will compare an intervention group to a waitlist control group to assess whether the intervention leads to increased guideline adherence.

Parents and Participants:

* Children will wear an accelerometer to track physical activity and sleep patterns.
* Parents will use a mobile app that delivers weekly lessons and behavior-related goals to encourage healthy movement behaviors in their children.
* Parents will complete questionnaires on their child's movement behaviors and development at baseline, 6 weeks, and 12 weeks.
* Additionally, children will undergo motor skills assessments, and parents will provide feedback on cognitive development and behavioral changes.

DETAILED DESCRIPTION:
The Shining Star study is a randomized controlled trial designed to evaluate the feasibility and preliminary effectiveness of a 12-week home-based mHealth intervention aimed at improving adherence to the 24-Hour Movement Guidelines (physical activity, sedentary behavior, and sleep) among preschool-aged children (3-4 years old). The trial consists of two groups: an intervention group receiving the mHealth intervention and a waitlist control group.

The primary objective is to determine if the intervention increases the proportion of children meeting all three 24-Hour Movement Guidelines. The intervention focuses on engaging parents through a mobile app, which delivers weekly lessons and behavior-related goals to promote healthy movement behaviors in children. Secondary objectives include assessing changes in child motor skills, cognition, behavioral problems and executive function, and BMI.

Study Design and Procedures:

Participants will be randomly assigned to either the intervention group or a waitlist control group. The intervention group will use the Shining Star mobile app, which provides short, weekly messages (less than 500 characters) and links to additional resources. The app will also include gamification elements, behavior trackers, and a forum for parents to connect with each other. Participants in the control group will receive access to the app after the 12-week intervention period.

Key measurements will be taken at three time points: baseline (Week 0), mid-point (Week 6), and at the end of the intervention (Week 12). Measurements include accelerometer data to assess physical activity, sedentary time, and sleep, anthropometrics to assess BMI, as well as parent-reported screen time, child motor skills, behavioral problems and executive function, and cognition. Usability and feasibility of the mobile app will be assessed through weekly app usage and feedback questionnaires.

Sample Size and Statistical Plan:

A total of 80 parent-child dyads (40 per group) will be enrolled in the study. A sample size of 30 families per group is expected to provide 80% power to detect a meaningful difference in the proportion of children meeting all three recommendations after 12 weeks. Based on a projected dropout rate of 25%, the target enrollment is 80 families.

Statistical analysis will focus on two primary hypotheses:

1. Whether a greater proportion of children in the intervention group meet the 24-Hour Movement Guidelines compared to the control group at 12 weeks.
2. Whether parents report that the intervention is feasible, with a target feasibility rating of ≥4.0/5.0 on a Likert scale.

Additional exploratory analyses will evaluate changes in child motor skills, behavioral problems, cognition, and growth as well as home-level and parent-level correlates.

Quality Assurance and Data Management:

Data will be collected using validated measures, and all data will be securely stored in REDCap. Clinical data collected at screening and follow-up visits, including accelerometer data and questionnaires, will be stored in a secure database at the University of Kansas Medical Center (KUMC). The data will undergo validation and consistency checks before analysis.

* Quality Assurance Plan: The research coordinator will ensure that accurate and complete data is transcribed from paper sources into REDCap. To maintain data quality, accuracy, and integrity, data entry will be performed twice. The REDCap data comparison tool will then be used to produce a final "Clean" entry.
* Missing Data Plan: Participants who do not complete the required assessments at baseline (Week 0), mid-point (Week 6), and end of the intervention (Week 12) will be excluded from the final analysis. Efforts will be made to retain participants throughout the study to minimize missing data.
* Statistical Analysis Plan: The primary analysis will compare the proportion of participants in the intervention and control groups meeting all three recommendations at 12 weeks using chi-square analysis. The secondary analysis will average the Likert scale responses across all weeks completed. Exploratory analyses will utilize linear regression to examine changes in outcomes between the treatment and control groups, along with iso-temporal substitution analysis to assess the impact of behavior substitution on child developmental outcomes. Additionally, the investigators will examine the relationship between meeting specific movement recommendations and child outcomes, with changes in theoretical components as potential mediators. Statistical significance will be set at p = 0.05 for analyses.

The study will also adhere to KUMC standard operating procedures for data collection, data analysis, and confidentiality as outlined in the study protocol.

ELIGIBILITY:
Inclusion (Child):

* Ages 3-4 years.
* Parent report that they meet 0 or 1 recommendation for physical activity, sleep, and screen-time as defined by the 24-hour movement guidelines. The physical activity recommendation is defined as greater than or equal to 3 hours/day of total physical activity, including 1 hour of moderate-to-vigorous physical activity. The sleep recommendation is defined as 10-13 hours/day. The sedentary behavior recommendation is defined as less than or equal to 1 hour/day of sedentary screen-time.

Inclusion (Parents):

* Parents must agree to use their mobile phone for the duration of the study (~12 weeks) and download the mobile app onto their phone.
* The parent/caregiver is fluent in English to participate in testing the mobile app.
* The parent/caregiver must be willing to travel to KUMC to complete study visits.

Exclusion (child):

* Mobility limitations as reported by the parent.
* Meeting two or more recommendations for physical activity, sleep, and screen-time.
* Sibling or household member is participating or participated in the study.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — male and female.
Enrollment: 80 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity (ActiGraph GT3X+ accelerometer) | Baseline, Week 6, and Week 12
  Physical activity will be device-measured using an ActiGraph GT3X+ accelerometer. Participants will wear the accelerometer on their wrist with a Velcro band for 14 consecutive days after their baseline visit, Week 6 visit, and Week 12 visit, removing it only for water-based activities (e.g., bathing).
Sleep (ActiGraph GT3X+ accelerometer) | Baseline, Week 6, and Week 12
  Sleep will be device-measured using an ActiGraph GT3X+ accelerometer. Participants will wear the accelerometer on their wrist with a Velcro band for 14 consecutive nights after their baseline visit, Week 6 visit, and Week 12 visit.
Screen Time | Baseline, Week 6, and Week 12
  Parents will report the average amount of time per day their child spent viewing screens (television, tablet, video game, cellphone, and other) while sitting or lying down, considering the past 30 days.
Feasibility and Acceptability of the Mobile App (Weekly Surveys) | Weekly
  Participant's randomized to the intervention will receive weekly surveys within the app to evaluate the feasibility and acceptability of the mobile health application. Parents will report how easy or difficult it was to achieve specific goals using a Likert scale ranging from 1 to 5, where 1 indicates a poor outcome and 5 indicates a better outcome.
Usability of the Mobile App (System Usability Scale) | Week 6 and Week 12
  Participants assigned to the intervention will rate their satisfaction with the app's design, appeal, and functionality using a 5-point Likert scale, which ranges from "Strongly Disagree" to "Strongly Agree." They will also complete the System Usability Scale (SUS), which also employs this 5-point Likert scale, at Week 6 and Week 12.

SECONDARY OUTCOMES:
Weight (kg) | Baseline, Week 6, and Week 12
  Weight will be measured in kg to the nearest 0.1 kg using a MX115 by BEFOUR scale.
Height (cm) | Baseline, Week 6, and Week 12
  Height will be measured in cm to the nearest 0.1 cm using a wall-mounted stadiometer.
BMI (kg/m²) | Baseline, Week 6, and Week 12
  Body mass index (BMI, kg/m²) will be calculated from the participant's collected height and weight measurements. These values will be combined to compute BMI, which will then be compared to national growth standards to determine the BMI z-score and categorize weight status (underweight, normal weight, overweight, or obesity).
Motor Skills - Grip Strength Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of upper extremity strength. Participants are asked to squeeze a Jamar® Plus+ Digital Hand Dynamometer as hard as they can, one hand at a time.
Motor Skills - 9-Hole Pegboard Dexterity Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of fine motor dexterity. Participants are asked to place 9 pegs into a Jamar® 9-Hole Peg Test Kit, then remove them as quickly as possible, one hand at a time.
Motor Skills - Standing Balance Test | Baseline, Week 6, and Week 12
  This NIH Toolbox assessment of balance involves participants performing a series of five progressively challenging poses on solid ground and a foam pad, with their eyes either open or closed. Each pose is held for 50 seconds, and postural sway is measured using an iPhone SE worn at the waist. Safety measures are in place to stop the test if necessary.
24-Hour Movement Behaviors | Week 6 and Week 12
  Parents will report updates to their child's average daily time spent on physical activity, nighttime sleep, and screen use during a typical week.
Motor Skills - 2-Minute Walk Endurance Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of cardiovascular endurance. Participants are asked to walk back and forth on a 50-foot course for two minutes, and the total distance walked is recorded in feet and inches.
Cognition - Picture Vocabulary Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of receptive vocabulary administered in a computer-adaptive test (CAT) format. Participants must choose which of four pictures best represents a word presented via audio.
Cognition - Flanker Inhibitory Control and Attention Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of inhibitory control and attention. The participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it.
Cognition - Dimensional Change Card Sort Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of cognitive flexibility and attention. The participant is asked to match a series of picture pairs to a target picture.
Cognition - Picture Sequence Memory Test | Baseline, Week 6, and Week 12
  An NIH Toolbox assessment of episodic memory. Participants are shown a number of activities, and then asked to reproduce the sequence of pictures as it was presented to them.
Behavioral Problems - BASC-3 | Baseline, Week 6, and Week 12
  The Behavior Assessment System for Children, Third Edition (BASC-3) is a tool that uses a Likert scale, specifically the "Never" to "Almost Always" scale, to assess behavioral problems in children. The scale ranges from 0 to 3, with 0 indicating "Never" and 3 indicating "Almost Always." Higher scores suggest greater behavioral problems, indicating a worse outcome.
Executive Function - BRIEF-P | Baseline, Week 6, and Week 12
  The Behavior Rating Inventory of Executive Function-Parent Version (BRIEF-P) is a tool that uses a Likert scale, "Never" to "Often," to assess executive function behaviors in preschool-aged children. Higher scores suggest greater difficulties with executive functioning, indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Chelsea L Kracht, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data will be submitted to the NICHD DASH database.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Data will be stored in the DASH data repository. Other requests for data and further information can be made to the PI, who will follow appropriate channels to distribute the data.

REFERENCES:
- [Derived] Kracht CL, Berge JM, LeBlanc M, Newton RL Jr, Rhodes RE, Bolamperti G, Snodgrass M, Redman LM. A Home-Based Intervention to Improve Adherence to the 24-Hour Movement Guidelines in Young Children: Protocol for a Mobile App-Based Randomized Control Trial. JMIR Res Protoc. 2026 Jan 29;15:e75621. doi: 10.2196/75621. PMID 41610419
- Available data/document: NIH Reporter Information — https://reporter.nih.gov/search/w2y2LWuI50aTEgDfuqR7lg/project-details/11017278 — Final Data set will be deposited into NICHD DASH database.